CLINICAL TRIAL: NCT00426686
Title: ADAMTS13-related Prognostic Factors in Adult and Pediatric Thrombotic Thrombocytopenic Purpura
Brief Title: ADAMTS13 in Thrombotic Thrombocytopenic Purpura
Acronym: ADAMTS13
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: PO51064
Record Dates: First submitted 2007-01-24; First posted 2007-01-25 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2011-04

CONDITIONS: Thrombotic Thrombocytopenic Purpura
Keywords: thrombotic thrombocytopenic purpura; prognostic factors; ADAMTS13
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples With DNA — March 2010
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Thrombotic thrombocytopenic purpura (TTP) is a thrombotic microangiopathy defined by the spontaneous formation of platelet thrombi in the microvessels. These platelet microthrombi are responsible for a mechanical hemolytic anemia, a thrombocytopenia and a multivisceral ischemia. TTP is a rare but life-threatening disease in the absence of appropriate treatment (PLASMATHERAPY). The onset of the disease usually occurs in adulthood (MOSCHCOVITZ syndrome) and rarely in childhood (UPSHAW-SCHULMAN syndrome). TTP is either sporadic or recurrent with multiple unpredictable relapses. TTP pathophysiology has remained obscure until a new metalloprotease, ADAMTS13, has been demonstrated to be involved in about 90% of all cases. Physiologically, ADAMTS13 function consists in limiting the size of von Willebrand factor (VWF) multimers and consequently, their hemostatic capacity. A large majority of TTP is associated with a severe deficiency of ADAMTS13. In most cases, ADAMTS13 severe deficiency is acquired via auto-antibodies to ADAMTS13; more rarely, ADAMTS13 deficiency is hereditary via ADAMTS13 gene mutations. ADAMTS13 auto-antibodies are either inhibitory of the catalytic activity or non inhibitory. ADAMTS13 mutations are spread all over the gene.

TTP prognosis is quite heterogeneous. Indeed, in about one third of the patients, TTP is refractory to PLASMATHERAPY and/or chronic relapsing. Until now, TTP prognosis factors are not known. Their identification is however crucial both to adapt the curative treatment of an acute episode (addition of first intention immunosuppressive agents to PLASMATHERAPY) and to prevent relapses.

In this context, the aim of the current project is to identify some ADAMTS13 related prognosis factors in TTP. A national prospective multicenter study including both adult and pediatric patients with TTP related to a severe ADAMTS13 deficiency will be designed over a three-year period. This study will involve our group as the French reference center for ADAMTS13 and 10 clinical departments from various French hospitals. Patients will be tested for ADAMTS13 activity and antigen, ADAMTS13 antibodies and ADAMTS13 gene sequencing. Our main hypothesis is that the inactivation of the ADAMTS13 domains crucial for its catalytic activity, either by inhibitory auto-antibodies (acquired TTP) or by genetic mutations (hereditary TTP) is a major bad prognosis factor.

DETAILED DESCRIPTION:
Thrombotic thrombocytopenic purpura (TTP) is a thrombotic microangiopathy defined by the spontaneous formation of platelet thrombi in the microvessels. These platelet microthrombi are responsible for a mechanical hemolytic anemia, a thrombocytopenia and a multivisceral ischemia. TTP is a rare but life-threatening disease in the absence of appropriate treatment (PLASMATHERAPY). The onset of the disease usually occurs in adulthood (MOSCHCOVITZ syndrome) and rarely in childhood (UPSHAW-SCHULMAN syndrome). TTP is either sporadic or recurrent with multiple unpredictable relapses. TTP pathophysiology has remained obscure until a new metalloprotease, ADAMTS13, has been demonstrated to be involved in about 90% of all cases. Physiologically, ADAMTS13 function consists in limiting the size of von WILLBRAND factor (VWF) multimers and consequently, their hemostatic capacity. A large majority of TTP is associated with a severe deficiency of ADAMTS13 activity leading to the accumulation of ultra large VWF multimers in plasma inducing the formation of platelet microthrombi in the microcirculation. In most cases, ADAMTS13 severe deficiency is acquired via auto-antibodies to ADAMTS13; more rarely, ADAMTS13 deficiency is hereditary via ADAMTS13 gene mutations. ADAMTS13 auto-antibodies are either inhibitory of the catalytic activity or non inhibitory. ADAMTS13 mutations are spread all over the gene.

TTP prognosis is quite heterogeneous. Indeed, in about one third of the patients, TTP is refractory to PLASMATHERAPY and/or chronic relapsing. Until now, TTP prognosis factors are not known. Their identification is however crucial both to adapt the curative treatment of an acute episode (addition of first intention immunosuppressive agents to PLASMATHERAPY) and to prevent relapses.

In this context, the aim of the current project is to identify some ADAMTS13 related prognosis factors in TTP. A national prospective multicenter study including both adult and pediatric patients with TTP related to a severe ADAMTS13 deficiency will be designed over a three-year period. This study will involve our group as the French reference center for ADAMTS13 and about 50 clinical departments from various French hospitals. Patients will be tested for ADAMTS13 activity and antigen, ADAMTS13 antibodies and ADAMTS13 gene sequencing. Our main hypothesis is that the inactivation of the ADAMTS13 domains crucial for its catalytic activity, either by inhibitory auto-antibodies (acquired TTP) or by genetic mutations (hereditary TTP) is a major bad prognosis factor.

ELIGIBILITY:
Inclusion Criteria:

* clinical suspicion of TTP
* Hemoglobin level < 10 g/dl (adult) or < 12 g/dl (child)
* Platelet level < 150 giga/l
* ADAMTS13 activity < 5%

Exclusion Criteria:

* Cancer
* Organ graft
* HIV infection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric patients with TTP related to a severe ADAMTS13 deficiency.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2006-11; Primary Completion 2009-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: paul COPPO, MD, PhD, Principal Investigator — Hôpital Saint Antoire, PARIS; Elie AZOULAY, MD, PhD, Study Director — Hôpital Saint Louis Paris; Benoît SCHLEMMER, MD, Study Director — Hôpital Saint Louis Paris; Eric OKSENHENDLER, MD, Study Director — Hôpital Saint Louis Paris; Fadi FAKHOURI, MD, Study Director — Hôpital Necker, PARIS; Jean-Paul MIRA, MD, PhD, Study Director — Hôpital Cochin, PARIS; Eric RONDEAU, MD, Study Director — Hôpital Tenon, PARIS; Jean-paul VERNANT, MD, Study Director — Hôpital la Pitié Salpétrière, PARIS; Nicolas SCHLEINITZ, MD, Study Director — CHU Conception, MARSEILLE; Gilles KAPLANSKI, MD, PhD, Study Director — CHU Conception, MARSEILLE; Albert BENSMAN, MD, Study Director — Hôpital Trousseau, PARIS; Chantal LOIRAT, MD, Study Director — Hôpital Robert Debré, PARIS; Brigitte BADER-MEUNIER, MD, Study Director — Hôpital Robert Debré, PARIS; Christophe PIGUET, MD, Study Director — Hôpital Dupuytren, LIMOGES; Guy PUTET, MD, Study Director — Hospices civils de LYON, LYON; Béatrice DUCOT, MD, Study Director — INSERM U569 Kremlin Bicêtre, Paris; Agnes VEYRADIER, MD, PhD, Study Director — Hôpital Antoine Béclère, CLAMART; Thierry LEBLANC, MD, Study Director — Hôpital Saint Louis Paris; Patrick NIAUDET, MD, PhD, Study Director — Hôpital Necker, PARIS; Christophe RIDEL, MD, Study Director — Hôpital Tenon, PARIS; Pascale POULLIN, MD, Study Director — CHU de la Conception, MARSEILLE; arlos FRANGIE, MD, Study Director — Hôpital Bicêtre, LE KREMLIN BICETRE; Hélène FRANCOIS, MD, Study Director — Hôpital Bicêtre, LE KREMLIN BICETRE; Olivier LAMBOTTE, MD, Study Director — Hôpital Bicêtre, LE KREMLIN BICETRE; Dominique BORDESSOULE, MD, PhD, Study Director — Hôpital Dupytren, LIMOGES; Stéphane GIRAULT, MD, Study Director — Hôpital Dupytren, LIMOGES; Hervé CHAMBOST, MD, Study Director — Hôpital de la Timone Enfants, Marseilles; Pierre BORDOGONI, MD, PhD, Study Director — Hôpital de Brabois-Hôpital d'Enfants, Vandoeuvre-lès-Nancy; Alexandra SALMON, MD, Study Director — Hôpital de Brabois- hôpital d'enfants, Vandoeuvre-lès-Nancy; Laurence CLEMENT, MD, Study Director — Hôpital de Brabois-Hôpital d'enfants, Vandoeuvre-lès-Nancy; Christian COMBE, MD, PhD, Study Director — Hôpital Pellegrin, Bordeaux; Sandrine MEUNIER, MD, Study Director — Hôpital Edouard Heriot, Lyon; Gwenaêlle ROUSSEY, MD, Study Director — Hôpital Hotel Dieu, Nantes; Mohammed HAMIDOU, MD, PhD, Study Director — Hôpital Hotel Dieu, Nantes; Bernard BONNOTTE, MD, PhD, Study Director — Hôpital du Bocage, Dijon; Yves TANTER, MD, Study Director — Hôpital du Bocage, Dijon; Jacques POURRAT, MD, PhD, Study Director — Hôpital de Rangueil, Toulouse; Marie-Christine THOURET, MD, Study Director — CHU de l'Archet 2, Nice; Philippe VANHILLE, MD, Study Director — CH de Valenciennes, Valenciennes; Nicolas LIMAL, MD, Study Director — Hôpital Henri Mondor, Créteil; Philippe REMY, MD, Study Director — Hôpital Henri Mondor, Créteil; Jean-Michel KORACH, MD, Study Director — CHG Châlons-en-Champagne, Châlons-en-Champagne; Carine GREIB, MD, Study Director — Hôpital Haut-Lévêque, Pesac; Jean-Louis PALLOT, MD, Study Director — CHI André Grégoire, Montreuil; Alain WYNCKEL, MD, Study Director — CHU de Reims, Reims; Claire CAZALETS, MD, Study Director — Hôpital Sud, Rennes; Bertrand DE CAGNY, MD, Study Director — CHU d'Amiens, Amiens; Claire PRESNE, MD, Study Director — CHU D'Amiens, Amiens; Cécile FOHRER, MD, Study Director — Hôpital de Haute-Pierre, Strasbourg; Karin BILGER, MD, Study Director — Hôpital de Haute-Pierre, Strasbourg; Bruno LIOURE, MD, Study Director — Hôpital de Haute-Pierre, Strasbourg; Raoul HERBRECHT, MD, PhD, Study Director — Hôpital de Haute-Pierre, Strasbourg; Dominique PLANTAZ, MD, PhD, Study Director — Hôpital Nord, Grenoble; Hubert NIVET, MD, PhD, Study Director — Hôpital Gatien de Clovheville, Tours; Emmanuel FLECK, MD, Study Director — Hôpital Saint Louis, La Rochelle; Jean-Philippe COINDRE, PH, Study Director — Centre Hospitalier du Mans, LE MANS; François MAURIER, PH, Study Director — Hôpital Sainte-Blandine Service de Médecine Interne, METZ; Mario OJEDA-URIBE, PH, Study Director — Centre Hospitalier Régional de MULHOUSE Hôpital Edouard Muller, Département d'Hématologie, Unité de thérapie cellulaire et greffes, MULHOUSE; Christophe RIDEL, PH, Study Director — Hôpital Tenon, Service de Néphrologie et de Transplantation rénale, PARIS; François BRIVET, PH, Study Director — Hôpital Antoine Béclère, Service de réanimation médicale, CLAMART; Sylvain LAVOUÉ, PH, Study Director — CHU Pontchaillou, Service de maladies infectieuses et réanimation médicale, RENNES; Sébastien CANET, PH, Study Director — Centre Hospitalier de Perpignan, Hôpital Saint-Jean, Service de Néphrologie, Hémodialyse, PERPIGNAN; François PROVOT, PH, Study Director — Centre Hospitalier Régional Universitaire de Lille, Hôpital Calmette, Pôle de Néphrologie, LILLE; Claude GUYOT, PH, Study Director — CHU de Nantes, Hôpital de jour et d'Hémodialyse pédiatrique; Xavier BELENFANT, PH, Study Director — CHI André Grégoire de Montreuil, Service de Néphrologie, Diabète et Dialyse, MONTREUIL; Laurent PERARD, PH, Study Director — Hôpital Edouard Herriot, Service de Médecine Interne, LYON; Edouard DEVAUD, PH, Study Director — CHR de Pontoise Hôpital René Dubos, Service de Médecine Interne- Néphrologie- Dialyse, PONTOISE; Arnaud BUFFIN, PH, Study Director — CH CHAMBERY, Service de Pédiatrie, CHAMBERY; Tarik KANOUNI, PH, Study Director — CHU Montpellier Hôpital Lapeyronie, Service d'Hématologie et Oncologie médicale, MONTPELLIER; Nicolas GAMBIER, PH, Study Director — Hôpital Avicenne, Service de Médecine Interne, BOBIGNY; Alain DEVIDAS, PH, Study Director — CH Sud-Francilien- Hôpital Gilles de Corbeil, Service d'Hématologie Clinique, CORBEIL-ESSONNES; Laure FEDERICI, PH, Study Director — CH Colmar- Hôpital Pasteur, Service de Médecine Interne, COLMAR; Michel FOULARD, PH, Study Director — CHRU de Lille- Hôpital Jeanne de Flandre, Service de Néphrologie pédiatrique, LILLE; Serge BOLOGNA, PH, Study Director — Hôpital Brabois Adulte, Service d'Hématologie, VANDOEUVRE-LÈS-NANCYS
Locations (1):
- Hôpital Antoine Béclère, Clamart, France

REFERENCES:
- [Background] Veyradier A, Obert B, Houllier A, Meyer D, Girma JP. Specific von Willebrand factor-cleaving protease in thrombotic microangiopathies: a study of 111 cases. Blood. 2001 Sep 15;98(6):1765-72. doi: 10.1182/blood.v98.6.1765. PMID 11535510
- [Background] Veyradier A, Obert B, Haddad E, Cloarec S, Nivet H, Foulard M, Lesure F, Delattre P, Lakhdari M, Meyer D, Girma JP, Loirat C. Severe deficiency of the specific von Willebrand factor-cleaving protease (ADAMTS 13) activity in a subgroup of children with atypical hemolytic uremic syndrome. J Pediatr. 2003 Mar;142(3):310-7. doi: 10.1067/mpd.2003.79. PMID 12640381
- [Background] Veyradier A, Lavergne JM, Ribba AS, Obert B, Loirat C, Meyer D, Girma JP. Ten candidate ADAMTS13 mutations in six French families with congenital thrombotic thrombocytopenic purpura (Upshaw-Schulman syndrome). J Thromb Haemost. 2004 Mar;2(3):424-9. doi: 10.1111/j.1538-7933.2004.00623.x. PMID 15009458
- [Background] Fakhouri F, Vernant JP, Veyradier A, Wolf M, Kaplanski G, Binaut R, Rieger M, Scheiflinger F, Poullin P, Deroure B, Delarue R, Lesavre P, Vanhille P, Hermine O, Remuzzi G, Grunfeld JP. Efficiency of curative and prophylactic treatment with rituximab in ADAMTS13-deficient thrombotic thrombocytopenic purpura: a study of 11 cases. Blood. 2005 Sep 15;106(6):1932-7. doi: 10.1182/blood-2005-03-0848. Epub 2005 Jun 2. PMID 15933059
- [Result] Ferrari S, Scheiflinger F, Rieger M, Mudde G, Wolf M, Coppo P, Girma JP, Azoulay E, Brun-Buisson C, Fakhouri F, Mira JP, Oksenhendler E, Poullin P, Rondeau E, Schleinitz N, Schlemmer B, Teboul JL, Vanhille P, Vernant JP, Meyer D, Veyradier A; French Clinical and Biological Network on Adult Thrombotic Microangiopathies. Prognostic value of anti-ADAMTS 13 antibody features (Ig isotype, titer, and inhibitory effect) in a cohort of 35 adult French patients undergoing a first episode of thrombotic microangiopathy with undetectable ADAMTS 13 activity. Blood. 2007 Apr 1;109(7):2815-22. doi: 10.1182/blood-2006-02-006064. PMID 17164349
- [Result] Malak S, Wolf M, Millot GA, Mariotte E, Veyradier A, Meynard JL, Korach JM, Malot S, Bussel A, Azoulay E, Boulanger E, Galicier L, Devaux E, Eschwege V, Gallien S, Adrie C, Schlemmer B, Rondeau E, Coppo P; Reseau d'Etude des Microangiopathies Thrombotiques (TMA-Rare Diseases Reference Center). Human immunodeficiency virus-associated thrombotic microangiopathies: clinical characteristics and outcome according to ADAMTS13 activity. Scand J Immunol. 2008 Sep;68(3):337-44. doi: 10.1111/j.1365-3083.2008.02143.x. PMID 18782260
- [Result] Loirat C, Girma JP, Desconclois C, Coppo P, Veyradier A. Thrombotic thrombocytopenic purpura related to severe ADAMTS13 deficiency in children. Pediatr Nephrol. 2009 Jan;24(1):19-29. doi: 10.1007/s00467-008-0863-5. Epub 2008 Jun 24. PMID 18574602
- [Result] Hommais A, Rayes J, Houllier A, Obert B, Legendre P, Veyradier A, Girma JP, Ribba AS. Molecular characterization of four ADAMTS13 mutations responsible for congenital thrombotic thrombocytopenic purpura (Upshaw-Schulman syndrome). Thromb Haemost. 2007 Sep;98(3):593-9. PMID 17849048
- [Derived] Weisinger J, Bouzid R, Fadlallah J, Provot F, Poullin P, Le Guern V, Ribes D, Martis N, Delmas Y, Chantepie S, Rieu V, Benhamou Y, Choukroun G, Marie M, Dana R, Veyradier A, Joly BS, Coppo P. Immune-mediated thrombotic thrombocytopenic purpura with systemic lupus erythematosus: clinical features and outcome. Lupus Sci Med. 2025 Jul 28;12(2):e001691. doi: 10.1136/lupus-2025-001691. PMID 40730415
- [Derived] Beranger N, Coppo P, Tsatsaris V, Boisseau P, Provot F, Delmas Y, Poullin P, Vanhoorelbeke K, Veyradier A, Joly BS. Management and follow-up of pregnancy-onset thrombotic thrombocytopenic purpura: the French experience. Blood Adv. 2024 Jan 9;8(1):183-193. doi: 10.1182/bloodadvances.2023011972. PMID 38039511
- [Derived] Beranger N, Tsatsaris V, Coppo P, Veyradier A, Joly BS. High sFlt-1 (Soluble fms-Like Tyrosine Kinase 1)/PlGF (Placental Growth Factor) Ratio in Pregnancy-Onset Thrombotic Thrombocytopenic Purpura. Hypertension. 2023 Sep;80(9):e140-e142. doi: 10.1161/HYPERTENSIONAHA.123.20987. Epub 2023 May 12. No abstract available. PMID 37170814
- [Derived] Joly BS, Stepanian A, Leblanc T, Hajage D, Chambost H, Harambat J, Fouyssac F, Guigonis V, Leverger G, Ulinski T, Kwon T, Loirat C, Coppo P, Veyradier A; French Reference Center for Thrombotic Microangiopathies. Child-onset and adolescent-onset acquired thrombotic thrombocytopenic purpura with severe ADAMTS13 deficiency: a cohort study of the French national registry for thrombotic microangiopathy. Lancet Haematol. 2016 Nov;3(11):e537-e546. doi: 10.1016/S2352-3026(16)30125-9. Epub 2016 Oct 3. PMID 27720178
- [Derived] Mariotte E, Azoulay E, Galicier L, Rondeau E, Zouiti F, Boisseau P, Poullin P, de Maistre E, Provot F, Delmas Y, Perez P, Benhamou Y, Stepanian A, Coppo P, Veyradier A; French Reference Center for Thrombotic Microangiopathies. Epidemiology and pathophysiology of adulthood-onset thrombotic microangiopathy with severe ADAMTS13 deficiency (thrombotic thrombocytopenic purpura): a cross-sectional analysis of the French national registry for thrombotic microangiopathy. Lancet Haematol. 2016 May;3(5):e237-45. doi: 10.1016/S2352-3026(16)30018-7. Epub 2016 Apr 16. PMID 27132698
- [Derived] Thouzeau S, Capdenat S, Stepanian A, Coppo P, Veyradier A. Evaluation of a commercial assay for ADAMTS13 activity measurement. Thromb Haemost. 2013 Oct;110(4):852-3. doi: 10.1160/TH13-05-0393. Epub 2013 Jul 11. No abstract available. PMID 23846249
- [Derived] Moatti-Cohen M, Garrec C, Wolf M, Boisseau P, Galicier L, Azoulay E, Stepanian A, Delmas Y, Rondeau E, Bezieau S, Coppo P, Veyradier A; French Reference Center for Thrombotic Microangiopathies. Unexpected frequency of Upshaw-Schulman syndrome in pregnancy-onset thrombotic thrombocytopenic purpura. Blood. 2012 Jun 14;119(24):5888-97. doi: 10.1182/blood-2012-02-408914. Epub 2012 Apr 30. PMID 22547583